CLINICAL TRIAL: NCT06815133
Title: Multicenter Retrospective Study on the Short- and Medium-Term Efficacy and Tolerance of Zilucoplan Therapy in a Cohort of French Patients With Anti-AChR Myasthenia Gravis
Brief Title: Effectiveness and Safety of Zilucoplan Treatment for French Patients With Myasthenia Gravis Over 3 Months
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Neuro01
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Anti-AChR Myasthenia Gravis treated with Zilucoplan
  Interventions: Drug: Zilbrysq

INTERVENTIONS:
Drug: Zilbrysq — Zilbrysq is a medicine used to treat generalized myasthenia gravis anti-AChR (a disease that leads to muscle weakness and tiredness) in adults whose immune system produces antibodies against a protein called the acetylcholine receptor. It is given as a subcutaneous injection (under the skin) once daily in a prefilled syringe that can be self-injected, and the dose depends on the patient's body weight. There are 3 available doses: 16.6 mg/0.416 mL for patients weighing less than 56 kg (123 lbs); 23 mg/0.574 mL for patients between 56 kg and less than 77 kg (123-170 lbs); and 32.4 mg/0.81 mL for patients weighing 77 kg and above (>170 lbs). This can be injected into the abdomen, front of the thighs, and back of the upper arms (only if administered by a caregiver),

SUMMARY:
This study called "Multicenter Retrospective Study on the Short- and Medium-Term Efficacy and Tolerance of Zilucoplan Therapy in a Cohort of French Patients with Anti-AChR Myasthenia Gravis", is investigating the effects of a new treatment called Zilucoplan (generic name: ZILBRYSQ) on patients in France with a condition known as myasthenia gravis. Myasthenia gravis is an autoimmune disease that causes muscle weakness that worsens throughout the day with activity and impacts the ability to work and perform daily activities. The study aims to see if Zilucoplan can improve muscle strength and quality of life over three months, while also assessing its tolerance and safety by monitoring side effects. Researchers hope this treatment will offer significant benefits for people with this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

- Confirmed diagnosis of myasthenia gravis with anti-AChR antibodies in patients treated with Zilucoplan

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from all the public hospitals in France where patients with confirmed myasthenia gravis with anti-AChR antibodies are given Zilucoplan as treatment under restricted access
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
MG-ADL scores | At the inclusion, at 1 month, at 3 months and at 6 months
  The MG-ADL is an 8-item patient-reported scale that measures myasthenia gravis symptoms and functional status. It assesses the impact of Myasthenia Gravis on the daily functions of the patients

SECONDARY OUTCOMES:
Garches scale scores | At the inclusion, at 1 month, at 3 months and at 6 months
  The Garches scale is a 9-item based on clinical examination which measures the severity of myasthenia symptoms and muscle function.
Evaluation of tolerance (M6) through the description of type of Adverse events | At 6 months
  Collect data on adverse events: total number of events, classification by type (mild, moderate, severe based on the " Common Terminology Criteria for Adverse Events (CTCAE) " scale)
Evaluation of tolerance (M6) through the description of the frequency of Adverse event | At 6 months
  number of adverse event per month
Adverse events possible association with the treatment (causality) | At 6 months
  causality (Certain / probable / possible / Unlikely / conditional / Unassessable)
Quality of life evaluation (MG-QoL15r) | At the inclusion, at 1 month, at 3 months and at 6 months
  Myasthenia gravis quality of life-15 revised (MG-QoL51r) is a 15-item quality of life scale designed to assess important aspects of the patient's experience related to myasthenia gravis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France